CLINICAL TRIAL: NCT04503993
Title: Utilizing Electronic Health Systems to Enhance Screening and Linkage to Care for Chronic Hepatitis B
Brief Title: Healthy Planet Hepatitis B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1423112
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Surface Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatitis B Healthy Planet Arm (Experimental): This is a single arm study where all patients eligible patients will receive a hepatitis B order set
  Interventions: Other: Hepatitis B surface antigen, Hepatitis B core antibody, and Hepatitis B surface antibody

INTERVENTIONS:
Other: Hepatitis B surface antigen, Hepatitis B core antibody, and Hepatitis B surface antibody — The hepatitis B tests are released into the electronic medical charts of at-risk patients who have never been screened for chronic hepatitis B using population health tools.

SUMMARY:
This quality improvement project utilizes Epic Health Planet to increase screening for chronic hepatitis B through the creation of registries and ordering of hepatitis B laboratory panels.

ELIGIBILITY:
Inclusion Criteria:

- Asian ancestry as determined by ethnicity/race, primary language, surname as recorded in the electronic health record

Exclusion Criteria:

- previously completed hepatitis B screening tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5004 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Completion of hepatitis B order panel | Within 1 year after placement of the order

SECONDARY OUTCOMES:
Linkage to care of those found to be infected with hepatitis B | Within 3 months after a positive HBsAg test

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No